CLINICAL TRIAL: NCT02500160
Title: Comparative Study of Total Knee Arthroplasty Using a Customized-patient Specific Instrument System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, KANG-IL KIM, professor & chairman, department of orthopaedic surgery, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMC 2011-058
Record Dates: First submitted 2015-07-13; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis, Knee; Arthroplasty, Replacement, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- patient specific instrumentation (MRI) (Experimental): MRI based patient-specific instrumentation
  Interventions: Device: Patient specific instrumentation (MRI)
- patient specific instrumentation (CT) (Active Comparator): CT based patient-specific instrumentation
  Interventions: Device: Patient specific instrumentation (CT)

INTERVENTIONS:
Device: Patient specific instrumentation (MRI)
  Arms: patient specific instrumentation (MRI)
Device: Patient specific instrumentation (CT)
  Arms: patient specific instrumentation (CT)

SUMMARY:
Patient-specific instrumentation (PSI) has been introduced in total knee arthroplasty (TKA) as a new technology for improving accuracy in restoration of the alignment and biomechanics of the lower limb. PSI in TKA refers to custom-made cutting jigs manufactured according to the patient's anatomic configuration of distal femur and proximal tibia based on preoperative magnetic resonance imaging (MRI) or computed tomography (CT) scans. MRI- and CT-based PSI systems are available from various manufacturers for preoperative planning. MRI offers precise visualization of articular cartilage without the risk of radiation exposure, but it is expensive and requires long scan times. In contrast, CT enables accurate identification of the contour of the femur and tibia at short scan times, but it does not provide information on the cartilage thickness and carries the risk of radiation exposure. As a result, there is a possibility of some discrepancy between the thickness of bone resection proposed by MRI- or CT-based PSI system and the actual thickness of bone cut. Although PSI has been the focus of study in many recent researches, there has been no clinical study comparing MRI-based and CT-based PSI systems in preoperative planning. Therefore the investigators questioned whether the MRI-based PSI that reflects the cartilage layer would provide more precision in TKA than the CT-based PSI. The purpose of this study was to investigate the accuracy of MRI-based PSI and CT-based PSI in predicting bone resection thickness in TKA.

ELIGIBILITY:
Inclusion Criteria:

* Of the patients who had been scheduled for TKA for the treatment of primary osteoarthritis only with varus deformity, those who had been waiting 6 weeks for TKA using an MRI-based or CT-based PSI system and had consented to the relatively new technique were enrolled in the study.

Exclusion Criteria:

* Patients with primary osteoarthritis with valgus deformity, rheumatoid arthritis, hemophilic arthritis, posttraumatic arthritis, other inflammatory arthritis, or a history of previous high tibial osteotomy were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The absolute differences (mm) between the planned resection thickness and the actual resection thickness in the femur and the tibia. | intraoperative time
  After bone resection using a patient-specific cutting jig, the actual thickness of resected bone was measured in 0.1 mm increments by the Vernier caliper (B.Braun-Aesculap, Tuttlingen, Germany) and compared with the planned resection thickness preoperatively using the PSI program.In the MRI group, the intraoperative cutting thickness was compared directly with the preoperatively planned thickness, whereas the presumed thickness of cartilage (2 mm) was added to actual thickness of resected bone from the lateral condyles in the CT group. Finally, the thickness of saw blade (1.27-mm) was added to every resected bone in all cases.

SECONDARY OUTCOMES:
radiographic assessment | postoperative 6 weeks
  The mechanical axis (MA) of the lower extremity and the coronal and sagittal alignments of the femoral and tibial components were measured on the anterior and lateral weight-bearing radiographs of the knee and the lower extremity orthogram before the surgery and 6 weeks after the surgery. The measurements were performed using a picture-acquiring communication system (PACS, Infinitt Healthcare, Seoul, Korea), and the data were recorded to one decimal place.

CONTACTS AND LOCATIONS:
Overall Officials: Kang-Il Kim, MD,PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea